CLINICAL TRIAL: NCT02894398
Title: Open-label, Multi-center, sINGlE Arm Clinical Study to Evaluate Efficacy/QoL in Women With HR+, HER2-, Regionally Recurrent or Metastatic Breast Cancer Receiving Palbociclib With an AI or Fulvestrant After Prior Endocrine Therapy
Brief Title: Study in Women With Advanced Breast Cancer Receiving Palbociclib With AI or Fulvestrant
Acronym: INGE-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iOM-04318
Record Dates: First submitted 2016-08-25; First posted 2016-09-09 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: HR+; HER2-; Locally advanced (inoperable or metastatic) Breast Cancer; Palbociclib; Aromatase inhibitor or fulvestrant; Pre-/perimenopausal receiving LHRH agonist / ovarian ablation; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Letrozole; Anastrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib+AI or Fulvestrant (Experimental): Letrozole as first-line or later line, Anastrozole as first-line, Exemestane as first-line, Fulvestrant as first-line or later line after prior endocrine therapy.
  Interventions: Drug: Palbociclib; Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Capsules (commercially available, obtained from local pharmacies), 125mg daily, 21 days, 7 days off, cycles of 28 days.
  Dose reductions: 100mg, 75mg (no change in administration schedule) Number of cycles: until disease progression, intolerable toxicity, death or any other reasons
  Other Names: Ibrance
Drug: Letrozole — Letrozole will be administered as basic therapy (commercially available tablets, obtained from local pharmacies) as followed: 2.5mg/daily, oral intake
  Other Names: Femara
Drug: Anastrozole — Anastrozole will be administered as basic therapy (commercially available tablets, obtained from local pharmacies) as followed: 1mg/daily, oral intake
  Other Names: Arimidex
Drug: Exemestane — Exemestane will be administered as basic therapy (commercially available tablets, obtained from local pharmacies) as followed: 25mg/daily, oral intake
  Other Names: Aromasin
Drug: Fulvestrant — Fulvestrant will be administered as basic therapy (commercially available injection, obtained from local pharmacies) as followed: 500mg/once monthly, intramuscular injection
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to evaluate the efficacy and quality of life in women with advanced breast cancer (locally advance inoperable or metastatic adenocarcinoma of the breast), HR+ / HER2-, who are treated with an aromatase inhibitor or fulvestrant as baseline therapy in combination with palbociclib (Ibrance)

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, single arm, non-comparative phase II study in women with HR+/HER2- advanced breast cancer receiving palbociclib in addition to an aromatase inhibitor or fulvestrant. The study will take place in Germany (85 study centers).

In total, 360 patients will be enrolled in this study. 6 treatment groups are planned. The study seeks to recruit 60 (58-62) patients per recruitment group. For first-line treatment with palbociclib - and letrozole (Enrollment Group 1), anastrozole (Enrollment Group 2), exemestane (Enrollment Group 3) or fulvestrant (Enrollment Group 4) and 60 (58-62) patients for second- or later-line treatment with palbociclib -and letrozole (Enrollment Group 5) or fulvestrant (Enrollment Group 6). Recruitment will be centrally monitored to allow closure of a respective group as soon as 60 (58-62) patients have been enrolled.

Treatment will be continued until disease progression, intolerable toxicity, death or any other reason. In case a combination partner is discontinued, palbociclib has to be discontinued. In case treatment with palbociclib is stopped, combination partner can be continued according to investigator's discretion. Irrespectively of the combination partner, the discontinuation of palbociclib is defined as end of treatment (EOT) in this study. After EOT the patient enters the follow-up period.

Primary end point is clinical benefit rate 24 weeks after the first study treatment of the patient.

A study independent, decentral, "virtual" biobank will be established. All patients will be asked to give consent for their tumor samples to be used for future investigational research. Study sites will inform the local pathologists about the patient's consent and ask for the tissue sample to be reserved for future analyses. The site is requested to collect contact details of the pathologist storing the tumor sample, the sample's identification number(s), and to document these in the eCRF.

The decision to perform subsequent investigational research studies on collected samples will be based on outcome data from this study or from new scientific findings related to the drug class or disease, as well as reagent and assay availability.

ELIGIBILITY:
Inclusion Criteria:

1. Personally signed written informed consent prior to beginning protocol specific procedures, including expected cooperation of the patient for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
2. Women with proven diagnosis of advanced, defined as locally advanced inoperable or metastatic, adenocarcinoma of the breast
3. Hormone-receptor-positive (HR+) disease, defined as estrogen-receptor-positive (ER+) and/or progesterone-receptor-positive (PgR+)
4. Human epidermal growth factor receptor 2-negative (HER2-) disease (HER2 neg/+ or HER2++ with CISH/FISH neg.)
5. Pre-/perimenopausal women receiving concomitant therapy with an luteinizing hormone-releasing hormone (LHRH) agonist / ovarian ablation or postmenopausal status
6. Age ≥18 years
7. Measurable disease as per Response Evaluation Criteria in Solid Tumors [RECIST] or bone-only disease
8. Patients scheduled for palliative treatment with an combination partner for first- or later-line
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
10. Adequate organ and marrow function
11. Resolution of all acute toxic effects of prior therapy, including radiotherapy Grade <1 (except toxicities not considered a safety risk for the patient) and recovery from surgical procedures
12. Fluent in spoken and written German

Exclusion Criteria:

1. Prior treatment with any CDK4/6 inhibitor
2. Prior adjuvant therapy with the respective endocrine combination partner if last intake <12 months prior to entering the study
3. Prior palliative therapy with the respective endocrine combination partner
4. More than one prior palliative chemotherapy
5. 5. Known hypersensitivity to letrozole, anastrozole, exemestane, fulvestrant or any of their excipients
6. Current use of food or drugs known to be potent inhibitors or inducers of CYP3A4 (refer to Appendix 15.4)
7. Current use of preparations containing St. John's Wort
8. Participation in other studies involving investigational drug(s) (Phases I-IV) within 2 weeks before the current study treatment begins
9. QTc > 480 msec on the screening ECG (using the QTcF formula and/or the QTcB (Bazett) formula); history of QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes
10. High cardiovascular risk, including, but not limited to recent myocardial infarction, severe/unstable angina and severe cardiac dysrhythmias in the past 6 months prior to enrollment
11. Patients with advanced symptomatic, visceral spread, that were at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement)
12. Diagnosis of any second malignancy within the last 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
13. Known, not-irradiated CNS metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 24 weeks after first administration of Palbociclib in combination with AI / fulvestrant
  CBR is defined as complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.

SECONDARY OUTCOMES:
Number of participants with Adverse Events as assessed by CTCAE V4.0 | From Date of Signed informed consent until PD, assessed up to 60 months.
  Adverse Events as characterized by type, frequency, severity (as graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v.4.03), and seriousness
Clinical Benefit Rate (CBR) | 48 weeks after first administration of Palbociclib in combination with AI / fulvestrant
  CBR is defined as complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.
Progression-free Survival rate | At 48 weeks (all patients) and 2 years (first-line patients only) after first administration of Palbociclib in combination with AI / fulvestrant
  Follow up 4 years after LPI
Overall Survival rate | At 48 weeks after first administration of Palbociclib in combination with AI / fulvestrant and yearly until EOS, assessed up to 60 months.
  Follow up 4 years after LPI
Time on treatment | From day of first treatment until permanent discontinuation (EOT), assessed up to 60 months.
  Study treatment will be continued until disease progression, intolerable toxicity, death or any other reason.
Dosage | From day of first treatment until EOT, assessed up to 60 months.
  * starting dose (mg)
  * adjusted doses (mg)
Adminstration schedule | From day of first treatment until EOT, assessed up to 60 months.
  - dates of administration
Health-related quality of life (QoL) | From date of signed informed consent until disease progression or start of next anti-cancer therapy: every 12 weeks, assessed up to 60 months.
  Health-related QoL will be assessed with the FACT-B (Functional Assessment of Cancer Therapy-Breast) questionnaire
Health-related fatigue | From date of signed informed consent until disease progression or start of next anti-cancer therapy: every 12 weeks, assessed up to 60 months.
  Fatigue will be assessed with the BFI (Brief Fatigue Inventory) questionnaire
Health-related anxiety and depression | From date of signed informed consent until disease progression or start of next anti-cancer therapy: every 12 weeks, assessed up to 60 months.
  Depression and anxiety will be assessed with the HADS-D (Hospital Anxiety and Depression Scale) questionnaire
Physician's assessment of patient's overall health status and change in health status compared to previous visit | From Screening until disease progression or start of next anti-cancer therapy, assessed up to 60 months.
  Assessed by 2 items at each cycle/at scheduled patient visit

CONTACTS AND LOCATIONS:
Overall Officials: iOMEDICO AG, Study Chair — Freiburg / Germany
Locations (70):
- Germany (70):
  - Research Site, Aachen
  - Research Site, Aschaffenburg
  - Augsburg
  - Research Site, Baden-Baden
  - Research Site, Berlin
  - Bochum
  - Bonn
  - Research Site, Bottrop
  - Bremerhaven
  - Research Site, Celle
  - Dessau
  - Research Site, Donauwörth
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Gerlingen
  - Goslar
  - Research Site, Göttingen
  - Göttingen
  - Greifswald
  - Güstrow
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hamburg
  - Homburg
  - Ilsede
  - Kaiserslautern
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Krefeld
  - Research Site, Langen
  - Research Site, Leer
  - Loerrach
  - Lübeck
  - Lüneburg
  - Mannheim
  - Minden
  - Research Site, Mönchengladbach
  - Research Site, Mühlhausen
  - Mülheim
  - Research Site, München
  - München
  - Research Site, Münster
  - Neumünster
  - Neuruppin
  - Offenburg
  - Oldenburg
  - Passau
  - Potsdam
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Rostock
  - Saarbrücken
  - Schorndorf
  - Research Site, Singen
  - Speyer
  - Stade
  - Stolberg
  - Stuttgart
  - Traunstein
  - Research Site, Ulm
  - Villingen-Schwenningen
  - Westerstede
  - Research Site, Wilhelmshaven
  - Witten
  - Würselen
  - Würzburg

IPD SHARING:
Plan to Share IPD: No